CLINICAL TRIAL: NCT02091414
Title: An Open Label Study to Evaluate the Effect of CellCept in Combination With Cyclosporine A and Steroids on Renal Function and the Prevention of Acute Rejection in Heart Transplant Patients.
Brief Title: A Study of CellCept (Mycophenolate Mofetil) in Combination Therapy in Heart Transplant Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20055
Record Dates: First submitted 2014-03-05; First posted 2014-03-19 (Estimated); Results first posted 2014-10-29 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Heart Transplantation
MeSH Terms: interventions — Mycophenolic Acid; Cyclosporine; Adrenal Cortex Hormones

ARMS (1):
- MMF, CsA, Corticosteroids (Experimental): Participants received mycophenolate mofetil (MMF) 1.0 grams (g), orally (PO), twice daily (BID) from within 24 hours of transplantation through Week 24. Participants also received an initial loading dose of cyclosporine A (CsA) 4 to 6 milligrams per kilogram (mg/kg) within 48 hours of transplantation, adjusted thereafter to a blood trough concentration of 150 to 300 nanograms per milliliter (ng/mL) through Week 24. Participants also received corticosteroids as per the practice of each participating center.
  Interventions: Drug: mycophenolate mofetil (MMF); Drug: cyclosporine A (CsA); Drug: corticosteroids

INTERVENTIONS:
Drug: mycophenolate mofetil (MMF) — 1.0 g PO BID
  Other Names: CellCept
Drug: cyclosporine A (CsA) — Initial loading dose of 4 to 6 mg/kg within 48 hours of transplantation, adjusted thereafter to a blood trough concentration of 150 to 300 ng/mL
Drug: corticosteroids — As per the practice of each participating center

SUMMARY:
This study will investigate the efficacy and safety of CellCept (1.5-2g/day po), in combination with a standard care regimen of cyclosporine A (trough level 150-200ng/mL) and steroids, in patients receiving a heart transplant. The anticipated time on study treatment is 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* patients receiving their first heart transplant (single organ transplant).

Exclusion Criteria:

* patients with a positive donor-specific cross-match at the time of transplantation;
* patients with any antibody-treated acute rejection;
* known contraindications to treatment with sirolimus;
* history of malignancy, other than excised non-melanoma skin cancer which has not recurred for 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (3):
- China (3):
  - Beijing
  - Fuzhou
  - Shanghai

RESULTS

PARTICIPANT FLOW:
Groups:
- Mycophenolate Mofetil (MMF) Plus (+) Cyclosporine A (CsA): Participants received MMF 1.0 grams (g), capsules orally (PO), twice daily (BID) from within 24 hours of transplantation through Week 24. Participants also received an initial loading dose of CsA 4 to 6 milligrams per kilogram (mg/kg) PO within 48 hours of transplantation, with dose adjustments thereafter as necessary to achieve a blood trough concentration of 150 to 300 nanograms per milliliter (ng/mL) through Week 24. Participants also received corticosteroids as per the practice of each participating center.
Period: Overall Study
Arm/Group | Mycophenolate Mofetil (MMF) Plus (+) Cyclosporine A (CsA)
Started | 36
Completed | 32
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: all enrolled participants who recieved at least 1 dose of study treatment.
Groups:
- MMF + CsA: Participants received MMF 1.0 g, capsules PO, BID from within 24 hours of transplantation through Week 24. Participants also received an initial loading dose of CsA 4 to 6 mg/kg PO within 48 hours of transplantation, with dose adjustments thereafter as necessary to achieve a blood trough concentration of 150 to 300 ng/mL through Week 24. Participants also received corticosteroids as per the practice of each participating center.
Arm/Group | MMF + CsA
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.83 (11.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Biopsy Proven Acute Rejection (BPAR) by Week
Description: Percentage of participants with BPAR of greater than or equal to (≥) International Society of Heart and Lung Transplant (ISHLT) Grade III. The ISHLT graded symptoms on a scale of Grade 0 through VI. Grade 0 equals (=) no rejection. Grade IA = regional (perivascular or interstitial) infiltration and no necrosis, and grade IB = dissemination but little infiltration and no necrosis. Grade II = 1 focus of invasive infiltration with or without (+/-) associated cardiomyocyte necrosis. Grade IIIA = 2 or more foci of invasive infiltration +/- associated cardiomyocyte necrosis, and grade IIIB = diffuse inflammatory pathological changes associated with cardiomyocyte necrosis. Grade IV = diffuse, infiltrative multi-foci +/- edema; +/- hemorrhage; and +/-vasculitis.
Time Frame: Day 1, Weeks 1, 2, 4, 8, 12, 16, 20 and 24
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MMF + CsA
Number analyzed (Participants) | 36
percentage of participants
  Day 1 | 0.0 [0.00 to 0.00]
  Week 1 | 0.0 [0.00 to 0.00]
  Week 2 | 2.78 [0.00 to 8.42]
  Week 4 | 2.78 [0.00 to 8.42]
  Week 8 | 2.78 [0.00 to 8.42]
  Week 12 | 2.78 [0.00 to 8.42]
  Week 16 | 2.78 [0.00 to 8.42]
  Week 20 | 2.78 [0.00 to 8.42]
  Week 24 | 2.78 [0.00 to 8.42]

2. Secondary Outcome: Percentage of Participants With Graft Loss Within 24 Weeks of Transplantation
Time Frame: Day 1, Weeks 1, 2, 4, 8, 12, 16, 20 and 24
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | MMF + CsA
Number analyzed (Participants) | 36
percentage of participants | 0.0

3. Secondary Outcome: Percentage of Participants Requiring Use of Additional Immunosuppressants Not Specified in the Protocol Within 24 Weeks of Transplantation
Time Frame: Day 1, Weeks 1, 2, 4, 8, 12, 16, 20 and 24
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | MMF + CsA
Number analyzed (Participants) | 36
percentage of participants | 0.0

4. Secondary Outcome: Percentage of Participants Discontinuing Immunosuppressants (MMF) for More Than 14 Consecutive Days or 30 Cumulative Days Within 24 Weeks of Transplantation
Time Frame: Day 1, Weeks 1, 2, 4, 8, 12, 16, 20 and 24
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MMF + CsA
Number analyzed (Participants) | 36
percentage of participants | 13.89 [2.02 to 25.76]

5. Secondary Outcome: Percentage of Participants Lost To Follow Up Within 24 Weeks of Transplantation
Time Frame: Day 1, Weeks 1, 2, 4, 8, 12, 16, 20 and 24
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | MMF + CsA
Number analyzed (Participants) | 36
percentage of participants | 0.0

6. Secondary Outcome: Percentage of Participants With Normal Serum Creatinine and Blood Urea Nitrogen (BUN) Values At Baseline (BL) And During Treatment
Time Frame: Day 1, Weeks 1, 2, 4, 8, 12, 16, 20 and 24
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | MMF + CsA
Number analyzed (Participants) | 36
percentage of participants
  Serum creatinine | 47.22
  BUN | 8.33

7. Secondary Outcome: Percentage of Participants With Normal Serum Creatinine and BUN Values at Baseline and Abnormal Values During Treatment
Time Frame: Day 1, Weeks 1, 2, 4, 8, 12, 16, 20 and 24
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | MMF + CsA
Number analyzed (Participants) | 36
percentage of participants
  Serum creatinine | 22.22
  BUN | 16.67

8. Secondary Outcome: Percentage of Participants With Abnormal Serum Creatinine and BUN Values at Baseline and Normal Values During Treatment
Time Frame: Day 1, Weeks 1, 2, 4, 8, 12, 16, 20 and 24
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | MMF + CsA
Number analyzed (Participants) | 36
percentage of participants
  Serum creatinine | 16.67
  BUN | 2.78

9. Secondary Outcome: Percentage of Participants With Abnormal Serum Creatinine and BUN Values at Baseline and During Treatment
Time Frame: Day 1, Weeks 1, 2, 4, 8, 12, 16, 20 and 24
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | MMF + CsA
Number analyzed (Participants) | 36
percentage of participants
  Serum creatinine | 13.89
  BUN | 72.22

ADVERSE EVENTS:
Time Frame: Adverse events were assessed at Day 1, and Weeks 1, 2, 4, 8, 12, 16, 20, and 24.
Description: All enrolled participants who received at least 1 dose of study drug were included in the safety analysis set.
Arm/Group | MMF + CsA
Serious Adverse Events (participants affected / at risk) | 2/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MMF + CsA (N=36)
Multiple organ failure (General disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MMF + CsA (N=36)
Rash (Skin and subcutaneous tissue disorders) | 1
Anemia (Blood and lymphatic system disorders) | 2
Wound complications (Injury, poisoning and procedural complications) | 2
Jaundice (Hepatobiliary disorders) | 2
Headache (Nervous system disorders) | 3
Epilepsy (Nervous system disorders) | 1
Lung infection (Infections and infestations) | 4
Folliculitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Impaired renal function (Renal and urinary disorders) | 6
Renal failure (Renal and urinary disorders) | 1
Insomnia (Psychiatric disorders) | 7
Dysphoria (Psychiatric disorders) | 4
Fever (General disorders) | 3
Impaired healing (General disorders) | 2
Elevated blood sugar (Investigations) | 14
Elevated blood lipids (Investigations) | 7
Elevated serum creatinine (Investigations) | 7
Elevated alanine aminotransferase (Investigations) | 7
Abnormal liver function tests (Investigations) | 7
Elevated serum bilirubin (Investigations) | 6
Leukocytosis (Investigations) | 6
Elevated aspartate aminotransferase (Investigations) | 5
High blood pressure (Investigations) | 2
Dyslipidemia (Investigations) | 1
Low blood pressure (Investigations) | 1
Increased platelet count (Investigations) | 1
Decreased serum glucose (Investigations) | 1
Increased serum albumin (Investigations) | 1
Increased heart rate (Investigations) | 1
Neutrophilic granulocytosis (Investigations) | 1
Elevated urea (Investigations) | 1
Positive anti hepatitis B antigen (Investigations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 17
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 14
Hyperlipidemia (Metabolism and nutrition disorders) | 4
Hypoproteinemia (Metabolism and nutrition disorders) | 1
Tachycardia (Cardiac disorders) | 8
Bradycardia (Cardiac disorders) | 3
Premature beat (Cardiac disorders) | 1
Palpitation (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 7
Indigestion (Gastrointestinal disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 2
Oral ulcers (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Hypertension (Vascular disorders) | 8
Wound bleeding (Vascular disorders) | 2
Thrombus (Vascular disorders) | 1
Perivenular inflammation (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.